CLINICAL TRIAL: NCT03024151
Title: The Effects of T4 Mono Replacement Versus T4/T3 Combination Replacement on Psychological Distress After Total Thyroidectomy in Thyroid Cancer Patients; Prospective, Randomized, Double Blind, T4 Comparative Clinical Study
Brief Title: The Effects of T4 Versus T4/T3 on Psychological Distress After Total Thyroidectomy in Thyroid Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: Dongnam Institute of Radiological & Medical Sciences (Other)
Responsible Party: Principal Investigator, Dongsik Bae, Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-05-010-001
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Thyroid Cancer; Distress; Depression; Anxiety; Fatigue
MeSH Terms: conditions — Thyroid Neoplasms; Depression; Anxiety Disorders; Fatigue | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T4/T3 combination replacement (Active Comparator): Comthyroid
  Interventions: Drug: Comthyroid
- T4 mono replacement (Active Comparator): Synthroid
  Interventions: Drug: Synthroid

INTERVENTIONS:
Drug: Comthyroid — T4/T3 combination replacement
  Arms: T4/T3 combination replacement
Drug: Synthroid — T4 mono replacement
  Arms: T4 mono replacement

SUMMARY:
The goal of this research is to compare the effects on psychological distress between T4 mono replacement group and T4/T3 combination replacement group after total thyroidectomy in thyroid cancer patients.

1. Subjects:

   * Psychologically distressed patients, such as depression, anxiety, and fatigue patient after total thyroidectomy with thyroid cancer are considered for participation. Screening of distress after total thyroidectomy is used HADS (Hospital Anxiety and Depression Scale) ≥ 8 for depression or anxiety, and MDASI-F (MD Anderson Symptom Inventory -Fatigue) ≥ 4 for fatigue.
2. Randomization:

   * Using the table of random sampling numbers, patients assign to T4 mono replacement group or T4/T3 combination replacement group.
3. Evaluation for distress:

   * Assessment will be made baseline, 4 weeks, 12 weeks and 24 weeks to investigate change of psychological distress (depression, anxiety, and fatigue). Level of distress after thyroidectomy will determine using Hospital Anxiety and Depression Scale (HADS), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI) for depression or anxiety, and Brief Fatigue Inventory (BFI) for fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who need thyroid hormone replacement therapy after total thyroidectomy for thyroid cancer
2. HADS (Hospital Anxiety and Depression Scale) ≥ 8 for depression or anxiety, or MDASI-F (MD Anderson Symptom Inventory -Fatigue) ≥ 4
3. Patient who maintain TSH recommendation range for TSH suppression according to ATA guidelines

Exclusion Criteria:

1. < 19 or ≥ 70 years old
2. Communication difficulties or inability to complete the necessary investigations and questionnaires
3. Inability to understand purpose of the study or disagree of participation
4. Past history of psychiatric treatment or diagnosis
5. Lactation or pregnancy
6. Past medical history of other cancer diagnosis or treatment
7. Any of severe comorbid medical conditions according to ASA score ≥ 3

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Psychological distress (depression or anxiety) assessed with HADS | baseline, 24 weeks
  Change from baseline HADS total score at 24 weeks
Fatigue assessed with MDASI-F | baseline, 24 weeks
  Change from baseline MDASI-F score at 24 weeks

SECONDARY OUTCOMES:
Depression assessed with BDI | baseline, 4, 12, 24 weeks
  Change from baseline BDI total score at 24 weeks
Anxiety assessed with BAI | baseline, 4, 12, 24 weeks
  Change from baseline BAI total score at 24 weeks
Fatigue assessed with BFI | baseline, 4, 12, 24 weeks
  Change from baseline BFI total score at 24 weeks
Response rate using BDI | baseline, 4, 12, 24 weeks
  improvement of depression sx. ≥ 50%
Response rate using BAI | baseline, 4, 12, 24 weeks
  improvement of anxiety sx. ≥ 50%
Response rate using BFI | baseline, 4, 12, 24 weeks
  improvement of fatigue sx. ≥ 50%
Remisssion rate using BDI | baseline, 4, 12, 24 weeks
Remission rate using BAI | baseline, 4, 12, 24 weeks
Remission rate using BFI | baseline, 4, 12, 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Dong sik Bae, Busan
  - Dongsik Bae, Busan